CLINICAL TRIAL: NCT01202383
Title: Household-based Chlorination of Drinking Water to Prevent Diarrhoeal Disease: a Randomized, Placebo-controlled Trial in India Using Sodium Dichloroisocyanurate (NaDCC) Tablets
Brief Title: Double-blinded Trial of Household-based Chlorination in India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Population Services International (Other); Partners for Affordable Technologies in Health (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); Chemical Council of America (Unknown); Medentech (Industry); Indian Institute of Health Management Research (Unknown)
Responsible Party: Principal Investigator, Thomas Clasen, Dr, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EH224
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Diarrhoea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NADCC tablets (Active Comparator)
  Interventions: Behavioral: Household-based water treatment with NADCC tablets
- Placebo tablets (Placebo Comparator)
  Interventions: Behavioral: Household-based water treatment with placebo tablets

INTERVENTIONS:
Behavioral: Household-based water treatment with NADCC tablets — Study participants will be supplied with tablets and encouraged to use them for treating their water daily
  Arms: NADCC tablets
Behavioral: Household-based water treatment with placebo tablets — Study participants will be supplied with tablets and encouraged to use them for treating their water daily
  Arms: Placebo tablets

SUMMARY:
The proposed study is a 12-month double-blinded, randomized, placebo-controlled trial to determine if the impact of treating water with chlorine at the household level is effective in preventing diarrhea among young children. For more than a century, chlorine has be used to treat water in municipal systems in developed countries. Lack of infrastructure has prevented its use in lower-income settings. NaDCC is a tablet form of chlorine that has been used for more than 30 years in emergencies and has recently been approved for routine treatment of drinking water by the WHO and US Environmental Protection Agency. The placebo will consist of the food-grade ingredients in the effective tablet, without the chlorine. Study participants will be supplied with tablets (intervention or placebo) and instructed to use the same to treat their water daily. Monthly follow-up visits will assess diarrhoea morbidity and weight-for-age Z scores in <5s. Chlorine residual and bacteriological quality of water stored in the home will be measured each month. The study will also assess the impact of the intervention on absenteeism from school and work and on health care expenditure for diarrhoea.

ELIGIBILITY:
Approximately 2000 households with children <5 will be enrolled.

Inclusion Criteria:

* Households with at least one child< 5
* Male and female head of household consent to participate
* Reside permanently in study area

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2163 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
diarrhoea morbidity | monthly visits for 12 months
  diarrhoea will be recorded among <5s and all ages

SECONDARY OUTCOMES:
weight for age Z-score | monthly visits for 12 months
  weight will be measured among <5s
bacteriological water quality in household storage container | monthly visits for 12 months
residual chlorine in household storage container | monthly visits for 12 months
absenteeism from school and work | monthly visits over 12 months
health care expenditure for diarrhea | One time visit

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Clasen, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Bhubaneswar, Odisha, India

REFERENCES:
- [Derived] Boisson S, Stevenson M, Shapiro L, Kumar V, Singh LP, Ward D, Clasen T. Effect of household-based drinking water chlorination on diarrhoea among children under five in Orissa, India: a double-blind randomised placebo-controlled trial. PLoS Med. 2013 Aug;10(8):e1001497. doi: 10.1371/journal.pmed.1001497. Epub 2013 Aug 20. PMID 23976883